CLINICAL TRIAL: NCT03815071
Title: Clinical Study of the Safety and Efficacy of Autologous Neural Stem Cells in the Treatment of Parkinson's Disease
Brief Title: A Study on the Treatment of Parkinson's Disease With Autologous Neural Stem Cells
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Allife Medical Science and Technology Co., Ltd. (Industry)
Collaborators: The First People's Hospital of Yunnan Province/First People's Hospital of Yunan Provinve New Kunhua Hospital (Unknown); Henan Provincial People's Hospital (Other); Beijing Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: NSC-PD-YNYY-01
Record Dates: First submitted 2019-01-21; First posted 2019-01-24 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ips-nsc treatment group (Experimental)
  Interventions: Drug: Ips-nsc cells

INTERVENTIONS:
Drug: Ips-nsc cells — Total dose of ips-nsc cells will be administered at day0.

SUMMARY:
This is a single center, single arm and open-label study to investigate the safety and efficacy of iPS-NCS with Parkinson's Disease

ELIGIBILITY:
Inclusion Criteria:

1. The subject is able to understand the research requirements, provide written informed consent, and complete the study in accordance with the procedures;
2. The subject is clearly diagnosed with Parkinson's;
3. Recorded disease progression over the past 6 months;
4. Vital organ function is satisfied: cardiac ultrasound indicates cardiac ejection fraction ≥ 50%, no obvious abnormality in ECG; blood oxygen saturation ≥ 90%; creatinine clearance calculated by Cockcroft-Gault formula ≥ 40ml/min; ALT and AST ≤ 3 times the normal range, total bilirubin ≤ 2.0 mg/dl;
5. Blood routine: Hgb≥80g/L, ANC≥1×109/L, PLT≥50×10/L;

Exclusion Criteria:

1. Mental illness or a neurological disease not associated with Parkinson's disease;
2. Serious other concomitant diseases (tumor, organ failure, etc.);
3. Subjects used a large amount of corticosteroids, immunoglobulins, immunosuppressants before entering the study;
4. Participated in other clinical trials of cell preparations and participated in other clinical trials within 3 months;
5. There are already cognitive impairments or depressions, etc., and the research cannot be completed well;
6. Female subjects who are breast-feeding or have a pregnancy plan recently.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-02-01 (Estimated); Primary Completion 2020-02-01 (Estimated); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
occurrence of treatment related adverse events | 1 year
  occurrence of treatment related adverse events that are possible, likely. Or definitely related to study treatment.

IPD SHARING:
Plan to Share IPD: No